CLINICAL TRIAL: NCT04677738
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Effects of a Bifidobacterium Breve Strain on Fat Loss in Healthy Adults
Brief Title: Investigation of the Effects of a Bifidobacterium Breve Strain on Fat Loss in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morinaga Milk Industry Co., LTD (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20BWHM
Record Dates: First submitted 2020-08-18; First posted 2020-12-21 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Overweight and Obesity
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo delivered in capsule format. Participants will be instructed to take 2 capsules of placebo for 4 weeks during the run-in period. On day 1 participants will be instructed to take 2 capsules of placebo in the morning before breakfast for 12 weeks.
  Interventions: Dietary Supplement: Placebo
- B. breve (Experimental): Capsule containing B breve strain. Participants will be instructed to take 2 capsules of placebo for 4 weeks during the run-in period. On day 1 participants will be instructed to take 2 capsules of B. breve strain in the morning before breakfast for 12 weeks.
  Interventions: Dietary Supplement: B. breve strain

INTERVENTIONS:
Dietary Supplement: B. breve strain — Probiotic capsule. Participants will be instructed to take 2 capsules of placebo for 4 weeks during the run-in period. On day 1 participants will be instructed to take 2 capsules of B. breve strain in the morning before breakfast for 12 weeks.
  Arms: B. breve
Dietary Supplement: Placebo — Placebo capsule. Participants will be instructed to take 2 capsules of placebo for 4 weeks during the run-in period. On day 1 participants will be instructed to take 2 capsules of placebo in the morning before breakfast for 12 weeks.
  Arms: Placebo

SUMMARY:
Overweight has become a critical issue in North America and the market value of weight loss products is expected to rise as the population becomes more health-conscious and aware of the risks associated with excess body weight. This randomized, placebo-controlled, clinical trial investigates the effect of Bifidobacterium breve supplementation with exercise intervention on fat loss.

DETAILED DESCRIPTION:
In early adulthood, excess body weight is a risk factor associated with several health complications later on in life and probiotics have been used for decades for maintaining intestinal health, and in recent years probiotics have been proposed for weight management. This randomized, placebo-controlled, clinical trial investigates the effect of Bifidobacterium breve supplementation with exercise intervention on fat loss.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 20 and 65 years of age, inclusive
* BMI from 25.0 to 29.9 kg/m2, inclusive
* Female participants are not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal (natural or surgically) for at least 1 year prior to screening
* Or, Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

  1. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
  2. Double-barrier method
  3. Intrauterine devices
  4. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
  5. Vasectomy of partner at least 6 months prior to screening
* Self-reported stable body weight for the past 3 months defined as not having gained or lost more than 5 kg of body weight throughout the 3 months prior to baseline
* Participants with the following body fat percentages as determined by Bioelectrical Impedance Analysis (BIA):

  1. Female: ≥ 30%
  2. Male: ≥ 20%
* Agrees to follow the diet and exercise guidelines for the duration of the study
* Willingness to complete questionnaires, records, and diaries associated with the study, to complete all clinic visits, and provide stool samples
* Provide voluntary, written, informed consent to participate in the study
* Healthy as determined by medical history, laboratory results and physical exam as assessed by the Qualified Investigator (QI)

Exclusion Criteria

* Women who are pregnant, breastfeeding or planning to become pregnant during the trial
* Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients
* Clinically significant abnormal laboratory results at screening as assessed by the QI
* Current or history of any significant gastrointestinal disease requiring medication (e.g. GERD, gastroenteritis)
* Irregular sleep schedule
* Chronic diarrhea or constipation
* Participants with hypertension and are on antihypertensive medication
* Type I or Type II diabetes
* Participants with hyperlipidemia and are on medication
* Self-reported sleep apnea
* Self-reported current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
* Unstable metabolic disease or chronic diseases as assessed by the QI
* History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom-free for 6 months
* Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case by case basis
* Major surgery in the past 3 months or individuals who have planned surgery during the trial period. Participants with minor surgery will be considered on a case-by-case basis by the QI
* Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
* Individuals with an autoimmune disease or are immune-compromised
* Self-reported HIV-, Hepatitis B- and/or C-positive diagnosis
* Blood/bleeding disorders as determined by laboratory results
* Self-reported mental or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation
* Metal implants that may affect the DXA scan results will be assessed on a case- by-case basis by the QI.
* Current use of prescribed medications listed in Section Prescribed Medications as follows:

  1. Beta-blockers and thiazide diuretics (within 4 weeks of baseline)
  2. Weight loss medication (within 4 weeks of baseline)
  3. Lipid-lowering medications (within 4 weeks of baseline)
  4. Anticoagulants and coagulants (within 4 weeks of baseline)
  5. Sleep medication
  6. Selective serotonin reuptake inhibitors (SSRI)
  7. Antibiotics
  8. Non-steroidal anti-inflammatory drugs (NSAIDs)
  9. Proton pump inhibitors (PPIs)
  10. Metformin (unless on a stable dose for the last 6 months)
* Current use of over-the-counter medications, supplements, foods and/or drinks as follows:

  1. OTC NSAIDs (PRN use is acceptable)
  2. OTC blood pressure medication or supplements (within 4 weeks of
  3. baseline)
  4. Lipid metabolising supplements (within 4 weeks of baseline)
  5. Fish oil and omega-3 supplements
  6. Red yeast rice
  7. Plant sterols and stanols
  8. OTC medication or supplements marketed for weight loss (within 4 weeks
  9. of baseline)
  10. Vitamin E supplements (within 4 weeks of baseline)
  11. Coagulant/anticoagulant supplements (within 4 weeks of baseline)
  12. PPIs
* Use of cannabinoid products within 60 days of baseline. History of cannabis used will be assessed on a case by case basis by the QI
* Use of tobacco products within 60 days of baseline
* Self-reported alcohol or drug abuse within the last 12 months
* High alcohol intake (average of > 2 standard drinks per day or > 10 per week)
* Current employment that calls for shift work or have worked shift work in the last 3 weeks
* Participation in other clinical research trials 30 days prior to screening
* Blood donation 30 days prior to screening, during the study, or a planned donation within 30-days of the last study visit
* Individuals who are unable to give informed consent
* Any other condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures, or which may pose a significant risk to the participant

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | B. Breve | Placebo
Started | 48 | 47
Completed | 44 | 45
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Population: for the ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | B. Breve | Placebo | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.71 (10.43) | 48.04 (11.16) | 44.84 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 43 | 43 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 1 | 0 | 1
  African American | 1 | 0 | 1
  Central American | 1 | 0 | 1
  East Asian | 3 | 0 | 3
  Eastern European White | 5 | 4 | 9
  Hispanic or Latino | 4 | 4 | 8
  Middle Eastern | 0 | 1 | 1
  Mixed | 0 | 1 | 1
  Other | 0 | 1 | 1
  South American | 1 | 0 | 1
  South Asian | 3 | 0 | 3
  South East Asian | 1 | 1 | 2
  Western European White | 28 | 35 | 63
Fat mass [Mean (Standard Deviation); unit: g] | 29587 (5942) | 30191 (4645) | 29886 (5320)
Fat mass ratio [Mean (Standard Deviation); unit: percentage of body weight] | 39.4 (7.5) | 40.5 (5.8) | 40.0 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat Loss (g)
Description: The difference in change in fat loss from baseline (g), as assessed by Dual-Energy X-Ray Absorptiometry (DXA), between B. breve and placebo after 12 weeks of supplementation. Body tissue density will be measured by a form of X-ray radiation and converted into body fat and muscle mass percentage for assessment
Time Frame: 12 weeks from baseline
Population: Per-protocol population after excluding the participants with concomitant medication or foods according to the judgement of principal investigator.
Measure: Mean (Standard Deviation); unit: g
Groups:
- B. Breve: Capsule containing B breve strain. Participants will be instructed to take 2 capsules of placebo for 4 weeks during the run-in period. On day 1 participants will be instructed to take 2 capsules of B. breve strain in the morning before breakfast for 12 weeks.
  B. breve: Probiotic capsule. Participants will be instructed to take 2 capsules of placebo for 4 weeks during the run-in period. On day 1 participants will be instructed to take 2 capsules of B. breve strain in the morning before breakfast for 12 weeks.
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
g | -78.38 (2186.66) | -9.43 (1428.19)

2. Primary Outcome: Change in Fat Loss (Percentage of Body Weight)
Description: The difference in change in fat loss from baseline (percentage of body weight), as assessed by Dual-Energy X-Ray Absorptiometry (DXA), between B. breve and placebo after 12 weeks of supplementation. Body tissue density will be measured by a form of X-ray radiation and converted into body fat and muscle mass percentage for assessment
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
percentage of body weight | -0.18 (2.01) | -0.12 (1.35)

3. Secondary Outcome: Body Weight
Description: The difference in change from baseline between B. breve and placebo in body weight after 12 weeks of supplementation
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
kg | -0.04 (2.45) | 0.10 (1.72)

4. Secondary Outcome: BMI
Description: The difference in change from baseline between B. breve and placebo in BMI after 12 weeks of supplementation
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
kilogram per square meter (kg/m^2) | -0.02 (0.90) | 0.03 (0.65)

5. Secondary Outcome: Android/Gynoid Fat Ratio
Description: The difference in change from baseline between B. breve and placebo in android/gynoid fat ratio as assessed by DXA after 12 weeks of supplementation. Android-gynoid percent fat ratio is a pattern of body fat distribution that is associated with an increased risk for metabolic syndrome in healthy adults.
  The measurement of android/gynoid fat ratio is defined as the ratio of the percentage of android fat to the percentage of gynoid fat.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of gynoid fat ratio
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
percentage of gynoid fat ratio | -0.02 (0.06) | 0.01 (0.06)

6. Secondary Outcome: Muscle Mass (g)
Description: The difference in change from baseline between B. breve and placebo in muscle mass (g) as assessed by DXA after 12 weeks of supplementation.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
g | 110.64 (1380.62) | 210.82 (1157.93)

7. Secondary Outcome: Muscle Mass (Percentage of Body Weight)
Description: The difference in change from baseline between B. breve and placebo in muscle mass (percentage of body weight) as assessed by DXA after 12 weeks of supplementation.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
percentage of body weight | 0.17 (2.04) | 0.15 (1.38)

8. Secondary Outcome: Waist Circumference
Description: The difference in change from baseline between B. breve and placebo in Waist circumference after 6 and 12 weeks of supplementation.
Time Frame: Baseline, 6 weeks and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
cm
  6 weeks from baseline | -0.22 (3.32) | -0.54 (3.31)
  12 weeks from baseline | -0.06 (2.92) | -0.54 (3.35)

9. Secondary Outcome: Hip Circumference
Description: The difference in change from baseline between B. breve and placebo in hip circumference after 6 and 12 weeks of supplementation.
Time Frame: Baseline, 6 weeks and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
cm
  6 weeks from baseline | -0.67 (3.97) | -0.80 (3.77)
  12 weeks from baseline | -1.04 (3.58) | -0.97 (4.51)

10. Secondary Outcome: Waist/Hip Circumference Ratio
Description: The difference in change from baseline between B. breve and placebo in waist/hip circumference ratio after 6 and 12 weeks of supplementation.
  The waist/hip circumference ratio is defined as the percentage of waist circumference to hip circumference. The change in waist/hip circumference ratio from baseline to week 12 was calculated.
Time Frame: Baseline, 6 weeks and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of hip circumference
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
percentage of hip circumference
  6 weeks from baseline | 0.00 (0.04) | 0.00 (0.05)
  12 weeks from baseline | 0.01 (0.04) | 0.00 (0.05)

11. Secondary Outcome: Microbiota Analysis: Shannon Index
Description: Alpha diversity at baseline and after 12-week intake were calculated by R. Alpha diversity index is usually unitless since it is a numerical value calculated by a mathematical formula, not a physical quantity.
  The Shannon Index (or Shannon-Wiener/Shannon-Weaver index) is a widely used metric in ecology to quantify alpha diversity, which measures both species richness and evenness.
  The value of the Shannon Index ranges from a minimum of zero, when there is only one species present (no diversity), to a maximum of ln(S), the natural logarithm of the total number of species (richness) to the base of Euler's number (e), which means all species are equally abundant. High values indicate a diverse, balanced community.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Shannon Index
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
Shannon Index
  Shannon@baseline | 5.92 (0.42) | 5.88 (0.52)
  Shannon@12 weeks | 6.00 (0.43) | 5.97 (0.50)

12. Secondary Outcome: Microbiota Analysis: Chao1 Index
Description: Alpha diversity at baseline and after 12-week intake were calculated by R. Alpha diversity index is usually unitless since it is a numerical value calculated by a mathematical formula, not a physical quantity.
  The Chao1 Index estimates total species richness, including rare/undetected species.
  The value of the Chao1 Index ranges from a minimum, close to zero (suggesting reduced richness, often observed in dysbiosis) to a theoretically unbounded maximum, as it depends on rare species. Higher values indicate greater estimated species richness, generally associated with a healthier gut microbiome, linked to resilience, metabolic versatility, and protection against pathogens.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Chao1 index
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
Chao1 index
  Chao1@baseline | 135.90 (31.16) | 141.50 (36.73)
  Chao1@12 weeks | 165.90 (40.57) | 158.20 (39.36)

13. Secondary Outcome: Microbiota Analysis: Evenness Index
Description: Alpha diversity at baseline and after 12-week intake were calculated by R. Alpha diversity index is usually unitless since it is a numerical value calculated by a mathematical formula, not a physical quantity.
  The Evenness Index measures how evenly individuals are distributed among species in a community, such as the gut microbiome. It complements species richness (the number of species) to describe diversity, ranging from 0 (only a single species, meaning there is no evenness.) to 1, where 1 indicates perfect evenness, meaning all species are equally abundant.
  Higher Evenness Index value (closer to 1) is generally considered better, as it suggests a more balanced and stable ecosystem. Conversely, lower value (closer to 0) is generally considered worse, as it suggests that a few species dominate the community, which can be associated with dysbiosis or an unhealthy gut microbiome.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Evenness Index
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
Evenness Index
  Evenness@baseline | 0.84 (0.026) | 0.84 (0.038)
  Evenness@12 weeks | 0.82 (0.030) | 0.82 (0.0058)

14. Secondary Outcome: Microbiota Analysis: Observed ASV Index
Description: Alpha diversity at baseline and after 12-week intake were calculated by R. Alpha diversity index is usually unitless since it is a numerical value calculated by a mathematical formula, not a physical quantity.
  Observed ASV (Amplicon Sequence Variants) Index refers to the number of distinct Amplicon Sequence Variants (ASVs) detected in a sample. ASVs are highly resolved sequences used to identify and differentiate microbial taxa, providing finer resolution than traditional Operational Taxonomic Units (OTUs).
  The range of Observed ASV Index in gut microbiome samples can range from a few hundred to several thousand, depending on several factors, including sample source, health status of the host, diet and lifestyle, as well as sequencing depth and methodology. Typically, higher Observed ASV Index indicates a more diverse microbial community, which can contribute to improved gut function and overall health.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Observed ASV Index
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
Observed ASV Index
  Observed ASV@baseline | 136.60 (32.94) | 132.40 (35.65)
  Observed ASV@12 weeks | 163.00 (38.68) | 156.1 (38.3)

15. Secondary Outcome: Microbiota Analysis: Faith's PD Index
Description: Alpha diversity at baseline and after 12-week intake were calculated by R. Alpha diversity index is usually unitless since it is a numerical value calculated by a mathematical formula, not a physical quantity.
  Faith's Phylogenetic Diversity (PD) is a measure used in ecology to quantify the biodiversity of a sample based on the phylogenetic tree. In the context of the gut microbiome, it specifically measures the diversity of microbial species by considering both the number of species present (richness) and the phylogenetic differences between them.
  In practice, the values can range from very low (close to zero, indicating low microbial diversity linked to various health issues) to very high (indicates greater evolutionary diversity, which may enhance ecosystem resilience and is generally considered better in the context of gut microbiome health.).
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Faith's PD Index
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
Faith's PD Index
  Faith's PD@baseline | 14.82 (3.17) | 14.57 (3.84)
  Faith's PD@12 weeks | 15.71 (3.81) | 15.53 (3.49)

16. Secondary Outcome: Change in Weight in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in weight in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Enterotype 1-B. Breve; Enterotype 1-Placebo: All subjects (regardless of B. breve or Placebo administration) are divided by enterotype. This sub-arm includes the subjects who share the same Enterotype 1, clustered at the genus level.
- Enterotype 2-B. Breve; Enterotype 2-Placebo: All subjects (regardless of B. breve or Placebo administration) are divided by enterotype. This sub-arm includes the subjects who share the same Enterotype 2, clustered at the genus level.
- Enterotype 3-B. Breve; Enterotype 3-Placebo: All subjects (regardless of B. breve or Placebo administration) are divided by enterotype. This sub-arm includes the subjects who share the same Enterotype 3, clustered at the genus level.
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
kg | -0.17 (2.76) | 0.46 (1.79) | 0.58 (1.96) | -0.25 (1.37) | -0.44 (1.93) | -0.77 (2.63)

17. Secondary Outcome: Change in Body Mass Index in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in body mass index in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
kilogram per square meter (kg/m^2) | -0.06 (1.04) | 0.16 (0.67) | 0.18 (0.6) | -0.11 (0.52) | -0.13 (0.7) | -0.3 (1.01)

18. Secondary Outcome: Change in Total Body Fat (g) in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in total body fat (g) in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
g | -238.24 (2301.91) | 55.77 (1290.03) | 31.8 (2251.64) | 51.67 (1506.94) | 335.14 (1883.4) | -793 (2325.77)

19. Secondary Outcome: Change in Total Body Fat (% of Body Weight) in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in total body fat (%) in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
percentage of body weight | -0.28 (2.02) | -0.14 (1.05) | -0.31 (2.26) | 0.09 (1.64) | 0.38 (1.79) | -1.02 (1.95)

20. Secondary Outcome: Change in Muscle Mass (g) in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in muscle mass (g) in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
g | 108.28 (1273.45) | 364.82 (981.21) | 600.4 (1660.45) | -82.87 (1441.46) | -580.57 (1202.31) | 550 (641.47)

21. Secondary Outcome: Change in Muscle Mass (% of Body Weight) in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in muscle mass (%) in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
percentage of body weight | 0.31 (2.04) | 0.2 (1.04) | 0.26 (2.28) | -0.12 (1.7) | -0.48 (1.86) | 1.18 (1.84)

22. Secondary Outcome: Change in Android Fat (g) in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in android fat (g) in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
g | -0.8 (269.1) | 83.14 (217.59) | -37.1 (411.6) | 1.13 (119.24) | -24.43 (190.81) | -122 (65.64)

23. Secondary Outcome: Change in Android Fat (% of Android Tissue) in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in android fat (%) in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of android tissue
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
percentage of android tissue | -0.56 (2.8) | 0.53 (1.17) | -0.84 (4.48) | 0.26 (1.92) | 0.33 (2.7) | -1.7 (0.87)

24. Secondary Outcome: Change in Gynoid Fat (g) in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in gynoid fat (g) in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
g | 83.52 (555.31) | 75.09 (310.83) | 94.50 (452.95) | -4.13 (524.2) | 107.29 (420.15) | 36 (677.02)

25. Secondary Outcome: Change in Gynoid Fat (% of Gynoid Tissue) in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in gynoid fat (%) in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of gynoid tissue
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
percentage of gynoid tissue | 0.2 (2.48) | 0.28 (1.75) | 0.74 (2.44) | 0.1 (2.65) | 0.36 (2.51) | -0.57 (1.6)

26. Secondary Outcome: Change in Android:Gynoid Fat Ratio in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in android:gynoid fat ratio in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of gynoid fat
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
percentage of gynoid fat | -0.01 (0.05) | 0.01 (0.06) | -0.04 (0.1) | 0.00 (0.06) | 0.02 (0.04) | -0.03 (0.02)

27. Secondary Outcome: Change in Waist Circumference in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in waist circumference in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
cm | -0.36 (3.46) | 0.00 (3.41) | 0.63 (2.38) | -0.94 (3.29) | 0.03 (0.93) | -2.4 (3.4)

28. Secondary Outcome: Change in Hip Circumference in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in hip circumference, in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
cm | -1.08 (4.08) | -0.26 (5.08) | -1.07 (3.3) | -1.77 (4.04) | -0.86 (2.13) | -2.1 (0.17)

29. Secondary Outcome: Change in Waist:Hip Circumference Ratio in Participant Groups Classified by Microbiota Composition at Week 0
Description: The change from baseline between B. breve and placebo in waist:hip circumference ratio in participant groups classified by microbiota composition at week 0, after 12 weeks of supplementation. These individual outcomes comprise relevant aspects of body composition. Each outcome will be analyzed separately and interpreted separately as well as collectively to inform relevant changes to body composition as a whole during the study.
Time Frame: 12 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of hip circumference
Arm/Group | Enterotype 1-B. Breve | Enterotype 1-Placebo | Enterotype 2-B. Breve | Enterotype 2-Placebo | Enterotype 3-B. Breve | Enterotype 3-Placebo
Number analyzed (Participants) | 25 | 22 | 10 | 15 | 7 | 3
percentage of hip circumference | 0.01 (0.05) | 0.00 (0.06) | 0.02 (0.04) | 0.01 (0.03) | 0.01 (0.01) | -0.01 (0.04)

30. Secondary Outcome: Total Cholesterol
Description: The difference in change from baseline between B. breve and placebo in total cholesterol after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
mmol/L | -0.05 (0.69) | 0.08 (0.53)

31. Secondary Outcome: HDL-cholesterol
Description: The difference in change from baseline between B. breve and placebo in HDL-cholesterol after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
mmol/L | -0.03 (0.18) | 0.00 (0.19)

32. Secondary Outcome: LDL-cholesterol
Description: The difference in change from baseline between B. breve and placebo in LDL-cholesterol after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
mmol/L | -0.06 (0.57) | 0.09 (0.47)

33. Secondary Outcome: Triglycerides
Description: The difference in change from baseline between B. breve and placebo in triglycerides after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
mmol/L | 0.09 (0.54) | -0.04 (0.50)

34. Secondary Outcome: Fasting Blood Glucose
Description: The difference in change from baseline between B. breve and placebo in fasting blood glucose after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
mmol/L | 0.05 (0.39) | 0.15 (0.33)

35. Secondary Outcome: HbA1c
Description: The difference in change from baseline between B. breve and placebo in HbA1c after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
percentage of glycated hemoglobin | 0.02 (0.17) | 0.03 (0.17)

36. Secondary Outcome: Fasting Insulin
Description: The difference in change from baseline between B. breve and placebo in fasting insulin after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
pmol/L | -9.43 (61.49) | 4.10 (28.25)

37. Secondary Outcome: Alkaline Phosphatase (ALP)
Description: The difference in change from baseline between B. breve and placebo in ALP after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
U/L | 2.83 (13.21) | 0.40 (8.44)

38. Secondary Outcome: Gamma-glutamyl Transferase (GGT)
Description: The difference in change from baseline between B. breve and placebo in GGT after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
U/L | 0.81 (5.58) | 0.25 (3.72)

39. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: The difference in change from baseline between B. breve and placebo in ALT after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
U/L | 0.60 (12.72) | -1.70 (7.63)

40. Secondary Outcome: Aspartate Transaminase (AST)
Description: The difference in change from baseline between B. breve and placebo in AST after 12 weeks of supplementation.
Time Frame: Baseline and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
U/L | 0.40 (5.91) | -1.77 (7.66)

41. Secondary Outcome: Frequency of Bowel Movements
Description: The difference in change from baseline between B. breve and placebo in Frequency of bowel movements after 6 and 12 weeks of supplementation.
Time Frame: Baseline, 6 and 12 weeks of supplementation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bowel movements
Arm/Group | B. Breve | Placebo
Number analyzed (Participants) | 42 | 40
bowel movements
  6 weeks from baseline | -0.36 (2.03) | 0.82 (2.68)
  12 weeks from baseline | -0.12 (2.05) | 0.62 (2.37)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | B. Breve | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 36/48 | 32/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B. Breve (N=48) | Placebo (N=47)
Abdominal discomfort (Gastrointestinal disorders) | 13 (18) | 10 (21) — Upset stomach, Nausea, Diarrhea, Vomiting, Constipation, Greenish stool, Heartburn, Indigestion, Ineffective straining at stool, Gastric pain
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (11) | 11 (17)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blood and urine biochemical indicator abnormal (Investigations) | 6 (6) | 0 (0) — Urinalysis abnormal NOS Alanine aminotransferase increased Urinalysis abnormal NOS Bilirubin total increased Urinalysis abnormal NOS Elevated K
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 12 (23) — Backache Muscle pain Pain in toe Plantar fasciitis Aching pain in hands, forearms, elbows Tenderness muscle Pain in hip
Arthropod sting, Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Bee sting Head injury
Pain, Fatigue, Pyrexia (General disorders) | 1 (1) | 3 (3) — Shooting pain Tiredness Chills & fever General body pain
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Mole changes
Headache (Nervous system disorders) | 18 (33) | 19 (47) — Headache Difficulty sleeping Sinus headache Tension headache
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Dysuria
Dysmenorrhea, Vulvovaginal discomfort (Reproductive system and breast disorders) | 2 (3) | 3 (6)
Oropharyngeal pain, Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) — Nose bleed Sore throat
Onychalgia, Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
none applicable

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT04677738/Prot_002.pdf
  • Statistical Analysis Plan (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04677738/SAP_003.pdf